CLINICAL TRIAL: NCT07035873
Title: Pediatric Cochlear Implant Remote Programming and Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Advanced Bionics (Industry)
Responsible Party: Principal Investigator, Ursula Findlen, Director of Audiology Research, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004526
Record Dates: First submitted 2025-05-22; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cochlear Implant Listeners
Keywords: pediatric; cochlear implant; remote programming; telehealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Remote Programming & Assessment (Experimental): Remote cochlear implant programming will be completed via the Advanced Bionics Remote Support iOS application. Remote assessment will be completed using the Advanced Bionics experimental Digital Audio Streaming (DAS) iOS application named EVA.
  Interventions: Behavioral: Remote Programming; Diagnostic Test: Remote Speech Perception

INTERVENTIONS:
Behavioral: Remote Programming — Use of the Advanced Bionics Target CI remote programming software to complete behavioral measurements of cochlear implant function and programming via telehealth.
Diagnostic Test: Remote Speech Perception — Use of digital audio streaming (DAS) through a proprietary platform to complete remote speech perception testing of performance with cochlear implants via telehealth.

SUMMARY:
This is a prospective, interventional study to evaluate efficacy and end user satisfaction of remote cochlear implant programming in the pediatric population. Additionally, this study will evaluate the long-term replicability of digital audio streaming (DAS) self-assessment speech perception measures via iOS mobile application.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the efficacy and end user satisfaction of mobile application based (1) remote cochlear implant programming and 2) self-administered audiological test measures in older children (13 to 20 year olds). Based on existing data, we hypothesize that remote programming is efficacious, and provides positive end user satisfaction. Additionally, while our prior work has shown that application-based speech perception outcomes are replicable when measured within one session, repeated testing over time may show learning effects.

ELIGIBILITY:
Inclusion Criteria:

* Cochlear implantation with an Advanced Bionics cochlear implant in at least one ear.
* At least 6 months post-implantation listening experience and at least 2 weeks of listening experience with Marvel cochlear implant external processor.
* Speech perception performance of at least 40% correct on standard of care speech perception measures in quiet for the ear to be used in the study
* Ages 13 years to 20 years, inclusive
* Ability and willingness to participate in remote programming sessions and self-administered assessment measures

Exclusion Criteria:

* Children under the age of 13
* Speech perception performance < 40% on SOC speech perception measures
* Cognitive or language deficits that preclude ability and willingness to participate in remote programming sessions and self-administered assessment measures, as identified by eMR diagnoses and the participant's primary clinical audiologist judgement.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and User Satisfaction- Participant | From enrollment to end of treatment at 6 months
  End user satisfaction as measured by survey of remote cochlear implant programming in the pediatric population. A variety of questions will be asked with Likert scale ratings, Scale = 1 (strongly disagree) to 5 (strongly agree), multiple choice, or open-ended questions.
Efficacy and User Satisfaction- Parent | From enrollment to end of treatment at 6 months
  End user satisfaction as measured by survey of remote cochlear implant programming in the pediatric population. A variety of questions will be asked with Likert scale ratings, Scale = 1 (strongly disagree) to 5 (strongly agree), multiple choice, or open-ended questions.

SECONDARY OUTCOMES:
DAS Speech Perception- Single Word Recognition | From enrollment to end of treatment at 6 months
  Speech perception performance measured via digital audio streaming (DAS) task via iOS application. Single word recognition is measured by typing the word heard and measured in percent correct.
DAS Speech Perception- Oldenburg Matrix Task | From enrollment to end of treatment at 6 months
  Speech perception performance measured via digital audio streaming (DAS) task via iOS application. The Oldenburg Matrix Task is a closed-set sentence in noise task in which the listener selects the five words heard in the sentence presented. Performance is measured in percent correct, speech recognition threshold (in dB), and signal-to-noise ratio slope.
DAS Speech Perception- Digits In Noise Task | From enrollment to end of treatment at 6 months
  Speech perception performance measured via digital audio streaming (DAS) task via iOS application. The Digits in Noise Task is a closed-set word in noise task in which the listener selects the three digits (numbers) heard. Performance is measured in percent correct and speech recognition threshold (in dB).
DAS Speech Perception- Soft Sound Detection | From enrollment to end of treatment at 6 months
  Speech perception performance measured via digital audio streaming (DAS) task via iOS application. The soft sound detection task is a threshold seeking tasks where the listener adjusts the level of a warble tone presented in noise until they deem it to be just barely noticeable. Performance is measured in dB level for frequencies 250, 500, 1000, 2000, 3000, 4000, and 6000 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula M Findlen, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States